CLINICAL TRIAL: NCT03750708
Title: Assessment of the Impact of the Use of the ARA 2 Connected Toothbrush on Short-term Oral Hygiene During the Pre-operative Period of Alveolar Bone Grafts for Patients With Unilateral or Bilateral Cleft Lip and Palate. Oral Hygiene and Connected Toothbrush Before Alveolar Bone Graft for Cleft Lip and Palate.
Brief Title: Oral Hygiene and Connected Toothbrush Before Alveolar Bone Graft for Cleft Lip and Palate
Acronym: HBD-GPP
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Unsuccessful study
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: APHP180025; 2018-A02062-53 (Registry Identifier: ID-RCB)
Record Dates: First submitted 2018-11-13; First posted 2018-11-23 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2022-11

CONDITIONS: Cleft Lip and Palate
Keywords: Alveolar bone graft complications, oral hygiene, cleft lip and palate, connected health
MeSH Terms: conditions — Cleft Lip

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ara® KOLIBREE toothbrush (Other): The Ara® KOLIBREE tooth brush is given to the child at the usual consultation one month before alveolar bone graft.
  Interventions: Device: Ara® KOLIBREE tooth brush
- Without Ara® KOLIBREE tooth brush (No Intervention): Usual consultation one month before alveolar bone graft.

INTERVENTIONS:
Device: Ara® KOLIBREE tooth brush — Use of the Ara® KOLIBREE tooth brush by the child one month before alveolar bone graft up to the time of surgery.
  The Ara® KOLIBREE tooth brush saves brush tracking data.
  Arms: Ara® KOLIBREE toothbrush

SUMMARY:
Alveolar bone graft is an essential step in the primary surgical treatment of unilateral or bilateral cleft lip and palate. The procedure involves repairing the alveolar cleft by an autologous iliac bone graft.

Clinical experience suggests that a large number of the post-operative complications in this procedure are related to pre-and post-operative oral hygiene issues.

The main objective of this research is the evaluation of pre-operative oral hygiene in children benefiting from alveolar bone graft and having a type Quad Helix orthodontic device.

The secondary objectives are to describe the use of the Ara ® Toothbrush by a population of children with a cleft lip and palate and to know whether the use of the Ara ® toothbrush has an influence on the occurrence of post-operative complications evaluated at 6 months of intervention (delays in scarring, suture dehiscence, fistulas, surgical site infections, total or partial graft loss).

DETAILED DESCRIPTION:
Alveolar bone graft is an essential step in the primary surgical treatment of unilateral or bilateral cleft lip and palate. The procedure involves repairing the alveolar cleft by an autologous iliac bone graft.

Clinical experience suggests that many post-operative complications in alveolar bone grafts are related to pre- and post-operative oral hygiene issues. This surgical procedure therefore requires optimal pre-and post-operative oral hygiene.

In addition, children with cleft lip and palate have a higher risk of oral hygiene issues, partly due to the systematic use of orthodontic devices such as Quad Helix.

Prevention of post-operative complications (delays in scarring, scar dehiscence, fistulas, infections of the surgical site, total or partial losses of the graft) requires patient education efforts in order to improve pre-operative oral hygiene.

Connected devices allow an objective follow-up tooth brushing and could be effective instruments in the primary and secondary prevention of pre-and post-operative complications linked to the alveolar bone graft, via a better oral hygiene.

Connected health is a growing and promising technology. It is important for physicians to demonstrate the efficiency of connected objects. Recent medico-economic studies have demonstrated the added value of connected devices as part of a general health monitoring, but more prospective assessments are required, especially in pediatric populations. Also, because of its importance in terms of public health, the field of oral hygiene is at the forefront of connected health applications.

The main objective of the research is the evaluation of pre-operative oral hygiene of children benefiting from an alveolar bone graft and having a type Quad Helix orthodontic device.

The secondary objectives are to describe the use of the Ara ® Toothbrush by a population of children with a cleft lip and palate and to know whether the use of the Ara ® toothbrush has an influence on the occurrence of post-operative complications evaluated at 6 months of intervention (delays in scarring, scar dehiscence, fistulas, surgical site infections, total or partial losses of the graft).

ELIGIBILITY:
Inclusion Criteria:

* Children aged 5 to 12 years.
* Children benefiting from iliac alveolar bone graft (first side for bilateral clefts) as part of the surgical management of unilateral a bilateral cleft lip and palate.
* Children benefiting from a pre-operative orthodontic treatment using Quad Helix type (usual protocol).
* Collection of the consent of the persons holding the parental authority and of the child participating in the study.
* Affiliation to social security.

Exclusion Criteria:

* Cognitive impairment preventing the satisfactory education for the use of the connected device.
* Chronic disease potentially favouring dental infections (congenital or acquired immunosuppression, congenital enamel disease).
* Children undergoing secondary alveolar bone grafts (after an unsatisfactory first alveolar bone graft) or undergoing surgery for the second side in bilateral clefts.
* Children participating in another interventional research.

Ages: 4 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2019-01-28 (Actual); Primary Completion 2021-02-28 (Actual); Study Completion 2021-02-28 (Actual)

PRIMARY OUTCOMES:
Oral hygiene score : CAO | Consultation 1 month before alveolar bone graft
  Individual CAO = C + A + O C : number of teeth decayed. A : number of teeth absent due to caries. O : number of teeth permanently blocked.
Oral hygiene score : CPITN | Consultation 1 month before alveolar bone graft
  CPITN : Community Periodontal Index of Treatment Needs : assessment of the periodontal status (index 0 (healthy) to 4).
Oral hygiene score : Silness-Löe Index | Consultation 1 month before alveolar bone graft
  Silness-Löe Index : index recording both soft debris and mineralized deposits on teeth (index 0 (no plaque) to 3).
Changes in oral hygiene score : CAO | Consultation 1 day before alveolar bone graft
  Individual CAO = C + A + O C : number of teeth decayed. A : number of teeth absent due to caries. O : number of teeth permanently blocked.
Changes in oral hygiene score : CPITN | Consultation 1 day before alveolar bone graft
  CPITN : Community Periodontal Index of Treatment Needs : assessment of the periodontal status (index 0 (healthy) to 4).
Changes in oral hygiene score : Silness-Löe Index | Consultation 1 day before alveolar bone graft
  Silness-Löe Index : index recording both soft debris and mineralized deposits on teeth (index 0 (no plaque) to 3).

SECONDARY OUTCOMES:
Description of the use of the Ara ® Toothbrush | Consultation at 1 day before alveolar bone graft
  Recorded data from the use of the Ara ® KOLIBREE tooth brush (Kolibree Pro interface)
Occurrence of post-operative complications | Consultation 6 months after alveolar bone graft
  Delays in scarring, scar dehiscence, fistulas, infections of the surgical site, total or partial losses of the graft

CONTACTS AND LOCATIONS:
Overall Officials: Roman Hossein Khonsari, MD PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hôpital Necker - Enfants Malades, Paris, France

IPD SHARING:
Plan to Share IPD: No